CLINICAL TRIAL: NCT05921968
Title: Evaluation of the Effect of Lactoferrin Versus Intravenous Iron Sucrose in Treatment of Iron Deficiency Anemia During Pregnancy
Brief Title: Effect of Lactoferrin Versus Intravenous Iron Sucrose in Treatment of Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amal A. Elkholy, lecturer of clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lactoferrin in Anemia
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Iron Deficiency Anemia
Keywords: Anemia in pregnancy; Lactoferrin; Iron Sucrose
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Pharmaceutical Preparations; Lactoferrin; Chemical Industry

STUDY DESIGN:
Intervention Model Description: prospective,randomized,open-label,parallel-group study
Masking Description: 100 opaque envelopes will be numbered serially and the corresponding letter which denotes the allocation will be put according to the electronic randomization table. Then all envelopes will be closed and put in one box. When the first patient arrives, the envelope will be opened and the patient will be allocated according to the letter inside
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Iron Sucrose group (Active Comparator): 50 pregnant women will receive 200 mg elemental iron in 100 ml 0.9 NaCl intravenous over 20 -30 minutes daily up to the total dose
  -The dose of the total iron sucrose to be administrated was calculated from the following formula: Total dose required = weight (kg) x (target Hb in g\dL - actual Hb in g\dL) x 2.4 + 500 mg rounded up to the nearest multiple of 100 mg
  Interventions: Drug: Intravenous iron sucrose
- Lactoferrin group (Active Comparator): 50 pregnant women will receive lactoferrin 100 twice daily orally .
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Intravenous iron sucrose — 200 mg elemental iron in 100 ml 0.9 NaCl intravenous over 20 -30 minutes daily up to the total dose)
  o The dose of the total iron sucrose to be administrated was calculated from the following formula: Total dose required = weight (kg) x (target Hb in g\dL - actual Hb in g\dL) x 2.4 + 500 mg rounded up to the nearest multiple of 100 mg
  Other Names: Intravenous iron sucrose(Sacrofer 100mg/5ml) was manufactured by Amoun company for pharmaceutical and chemical industry ,Egypt.
  Arms: Intravenous Iron Sucrose group
Drug: Lactoferrin — 100 mg twice daily orally before breakfast and dinner
  Other Names: lactoferrin 100 mg (Pravotin100 mg sachet)was manufactured by Hygint company for pharmaceutical and chemical industry,Egypt. Egypt) twice daily orally .
  Arms: Lactoferrin group

SUMMARY:
Iron deficiency is the most common nutritional deficiency and the most common cause of anemia. Anemia has a significant impact on the health of the fetus as well as that of the mother. It impairs the oxygen delivery through the placenta to the fetus and interferes with the normal intrauterine growth, leading to fetal loss and perinatal deaths. Anemia is associated with increased preterm labor (28.2%), preeclampsia (31.2%), and maternal sepsis.

The study aims to compare the effect of Lactoferrin versus intravenous iron sucrose for the treatment of iron deficiency anemia during pregnancy.

DETAILED DESCRIPTION:
Iron deficiency is the most common nutritional deficiency and the most common cause of anemia. Anemia has a significant impact on the health of the fetus as well as that of the mother. It impairs the oxygen delivery through the placenta to the fetus and interferes with the normal intrauterine growth, leading to fetal loss and perinatal deaths. Anemia is associated with increased preterm labor (28.2%), preeclampsia (31.2%), and maternal sepsis.

The study aims to compare the effect of Lactoferrin versus intravenous iron sucrose for the treatment of iron deficiency anemia during pregnancy.

The study will include 100 pregnant women with moderate iron deficiency anemia. They will assigned randomly in to 2 groups. Each group will contain 50 patients.

The first group will receive intravenous iron sucrose (sacrofer 100mg/5ml)as 200 mg elemental iron in 100 ml 0.9 NaCl over 20-30 minutes up to the total dose -Total dose will be calculated from this equation=weight(kg)x(target Hb in g/dl-actual Hb in g/dl)x2.4+500 rounded up to the nearest multiple of 100 mg The second group will receive lactoferrin 100 mg twice daily orally before breakfast and before dinner (pravotin 100 mg sachets will be dissolved in ¼ glass of water). Patients will be advised to avoid coffee, milk products and antacid before and after the dose of lactoferrin.

1. Baseline assessment:

All women in the study will be submitted to:

1. Complete History Taking Including:

   * Personal history: This included name, age, duration of marriage, last menstrual period, parity, occupation and special habits.
   * 1st day of last menstrual period.
   * Estimated gestational age
   * Contraceptive history
   * Obstetric history Including:
   * Full details of previous pregnancies (Date, outcome, onset and mode of delivery, gestational age at delivery and any associated complication or history of similar disorder, spacing between each pregnancy.
2. General Examination Included: Weight, height, body Mass Index (BMI), temperature, pulse, blood pressure, chest and cardiac examination, signs of anemia
3. Abdominal Examination
4. Fetal monitoring: To confirm fetal maturity and fetal wellbeing by non-stress test and biophysical profile.
5. U/S investigation: To confirm gestational age and exclude associated congenital anomalies.

Investigations:

* Complete blood sample (CBC), total iron binding capacity and Transferrin saturation will be done in Ain Shams Maternity Hospital Labs.
* Serum ferritin will be sent to any private lab.
* Kidney function tests and liver function tests. 2. Follow up assessment:

  * Anemic pregnant women will be followed up every 4 weeks until delivery.
  * In between visits, patients will be contacted via phone for monitoring of any side effects.

    3. End of study assessment:
* the same laboratory tests will be done with monitoring of any signs or symptoms of anemia until Hb level > 11 g/dl

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with iron deficiency anemia.
* Microcytic hypochromic anemia, moderate anemia (Hb 8 to 9.9 g/dl) and S. Ferritin levels <12 ng/dl as per WHO guidelines
* Gestational age: - 13-26 weeks.
* Singleton viable pregnancy
* Lastly, agreement to participate and sign the informed consent was a basic prerequisite

Exclusion Criteria:-

* Women with a history of anemia due to any other causes such as chronic blood loss, hemolytic anemia, and thalassemia (including thalassemia trait).
* Severe anemia <7 g/dl requiring blood transfusion, bronchial asthma, clinical and/or laboratory evidence of hepatic, renal, hematologic or cardiovascular abnormalities.
* History of peptic ulcer.
* Hypersensitivity to iron preparations and treatment with any other iron preparation in the last one month before study entry.
* Suspected acute infection.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the effect of oral lactoferrin as compared to intravenous iron sucrose on the serum level of ferritin | 4 weeks
  estimation serum ferritin level
evaluate the effect of oral lactoferrin as compared to intravenous iron sucrose on the serum level of hemoglobin | 4 weeks
  estimation hemoglobin level

SECONDARY OUTCOMES:
evaluation of lactoferrin side effect | 4 weeks
  assessment of the incidence rate of nausea, vomiting and GIT upset
the incidence rate of constipation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Sabri, professor, Study Chair — Department of Clinical Pharmacy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Artym J, Zimecki M, Kruzel ML. Lactoferrin for Prevention and Treatment of Anemia and Inflammation in Pregnant Women: A Comprehensive Review. Biomedicines. 2021 Jul 27;9(8):898. doi: 10.3390/biomedicines9080898. PMID 34440102